CLINICAL TRIAL: NCT02063139
Title: A Single (Assessor)-Blind, Randomised, Three-period, Cross-over Study to Compare the Safety of Flutiform pMDI, Fluticasone pMDI, and Beclometasone Autohaler in Paediatric Subjects Aged 5 to Less Than 12 Years With Mild Persistent Asthma by Means of Knemometry
Brief Title: Knemometry Study to Compare the Systemic Safety of Flutiform pMDI, Fluticasone pMDI and Beclometasone Autohaler in Paediatric Subjects Aged 5 to Less Than 12 Years.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mundipharma Research Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: FLT2504; 2013-004719-32 (EudraCT Number)
Record Dates: First submitted 2014-02-11; First posted 2014-02-14 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Mild Persistent Asthma
Keywords: Knemometry
MeSH Terms: interventions — fluticasone-formoterol; Fluticasone

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- Flutiform 50/5 ug (2 puffs bid) pMDI (Experimental): Flutiform 50/5 ug (2 puffs bid) pMDI
  Interventions: Drug: Flutiform 50/5 ug (2 puffs bid) pMDI
- Fluticasone 50 ug (2puffs bid) pMDI (Active Comparator): Fluticasone 50 ug (2puffs bid) pMDI
  Interventions: Drug: Fluticasone 50 ug (2puffs bid) pMDI
- Beclometasone Autohaler 50 ug (2 puffs bid) (Other): Active control
  Interventions: Drug: Beclometasone Autohaler 50 ug (2 puffs bid)

INTERVENTIONS:
Drug: Flutiform 50/5 ug (2 puffs bid) pMDI
  Arms: Flutiform 50/5 ug (2 puffs bid) pMDI
Drug: Fluticasone 50 ug (2puffs bid) pMDI
  Arms: Fluticasone 50 ug (2puffs bid) pMDI
Drug: Beclometasone Autohaler 50 ug (2 puffs bid)
  Arms: Beclometasone Autohaler 50 ug (2 puffs bid)

SUMMARY:
Aim of the study is to investigate the short-term growth in children with asthma aged 5-11 years in treatment with fluticasone propionate / formoterol spray (flutiform®) 200/20 micrograms per day

ELIGIBILITY:
Inclusion Criteria

Subjects to be included in the study are those who meet all of the following criteria:

1. Male and Female subjects 5 to <12 years old. Female subjects must be pre-menarche to be eligible.
2. Subjects must be pre-adolescent without any signs of puberty (acc. to Tanner scale).
3. Subjects are in normal range for their age in height and weight. Weight and height measurements should fall within the percentile range 3-97-% of normal values for age according to Danish growth charts.
4. Known history of mild intermittent or persistent reversible asthma for ≥ 3 months prior to the screening visit.
5. Require:

   1. only inhaled SABA therapy (e.g. Bricanyl Turbuhaler) on an as required basis, and/or
   2. Regular non-ICS controller medications for asthma (e.g., cromones or leukotriene receptor antagonists) at a stable dose for ≥ 3 months prior to the screening visit.
6. No ICS for >2 weeks prior to the screening visit.
7. Demonstrates adequate spirometry technique and able to use a home PEFR meter.
8. Demonstrated FEV1 of ≥ 80% predicted value at visit 1following appropriate withholding of asthma medications (if applicable) (no SABA use within 6 hours of the PFT).
9. Demonstrated satisfactory technique in the use of the pMDI plus spacer and Autohaler devices.
10. Must be continent of urine and willing to perform (with parental/guardian help) overnight urine collections.
11. Willing and able to complete morning and evening PEFR measures with the help of a parent or guardian, if necessary, and attend all study visits.
12. Willing and able to substitute pre-study prescribed inhaled asthma medication for the entire duration of the study with study medication.
13. Written informed consent obtained as per national laws.

    Inclusion Criteria required following run-in:
14. FEV1 within ≤20% of the visit 1 value following appropriate withholding of rescue medication (no salbutamol Airomir Autohaler use within 6 hours of the PFT).

Rescue medication use on ≤2 days during the last 7 days of the run in period. Exclusion Criteria

Subjects to be excluded from the study are those who meet any of the following criteria:

1. Require medications other than inhaled SABAs and/or regular non-ICS controller medications (e.g., cromones or leukotriene receptor antagonists) to maintain asthma control.
2. ICS use within ≤ 2 weeks prior to the screening visit.
3. Any asthma exacerbation of any severity for at least 3 months prior to the screening visit.
4. Any fracture in the leg to be measured by knemometry ≤6 months prior to the screening visit.
5. Any metabolic disorders or other diseases that may impact on normal growth patterns.
6. Near fatal or life-threatening asthma within the past year.
7. Hospitalisation or an emergency visit for asthma within the past 6 months.
8. History of oral or injectable corticosteroid medication ≤3 months prior to the screening visit.
9. Evidence of a clinically unstable disease, as determined by medical history, clinical laboratory tests, and physical examination that, in the Investigator's opinion, preclude entry into the study. "Clinically significant" is defined as any disease that, in the opinion of the Investigator, would put the subject at risk through study participation, or which would affect the outcome of the study.
10. No major surgery requiring general anesthesia for at least 3 months prior to the screening visit.
11. No febrile illnesses with temperature > 39°C within a week of the screening visit.
12. In the Investigator's opinion a clinically significant upper or lower respiratory infection within 4 weeks prior to the screening visit.
13. Significant, non-reversible active pulmonary disease (e.g. cystic fibrosis, bronchiectasis, tuberculosis).
14. Subjects who have taken β- blocking agents, tricyclic antidepressants, monoamine oxidase inhibitors, astemizole (Hismanal), quinidine type antiarrythmics, or potent CYP 3A4 inhibitors such as ketoconazole within 1 week prior to the screening visit.
15. Current use of medications, other than those allowed in the protocol.
16. Current evidence of hypersensitivity or idiosyncratic reaction to test medications or components.
17. Receipt of an Investigational medicinal product within 30 days of the screening visit.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2014-02; Primary Completion 2014-06 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
To show non-inferiority of flutiform pMDI 50/5 µg (2 puffs bid) versus fluticasone pMDI 50 µg (2 puffs bid) based on the mean lower leg growth rates. | Change from baseline in growth rate during the each treatment and washout period which is 2 weeks
  Lower leg length will be measured in the afternoon, between 13:00 and 19:00h. Each individual subject will have their knemometry measurements performed at the same time of day (+/- 1 hour).

SECONDARY OUTCOMES:
To compare the safety of flutiform pMDI 50/5 µg (2 puffs bid) versus fluticasone pMDI 50 µg based on overnight urinary free cortisol (corrected for creatinine). | every two weeks for duration of study which is two months.
  Subjects will empty their bladder into the toilet before going to bed at night (or no later than at 10pm). This urine will not be collected. This voiding time will be recorded as the start time of the urine collection. Urine passed after this time during the night (if any) and until 8 am in the morning will be collected into a clean container. Subjects will empty their bladders a final time at 8 am in to the container. This voiding time will be recorded as the stop time of the urine collection.

CONTACTS AND LOCATIONS:
Locations (1):
- Asthma and Allergy Children's Clinic, Randers, Denmark

REFERENCES:
- [Derived] Wolthers OD, Mersmann S, Dissanayake S. A Pilot Study of the Normative Range of Overnight Urinary Free Cortisol Corrected for Creatinine in Children. Clin Drug Investig. 2018 Apr;38(4):313-318. doi: 10.1007/s40261-017-0609-x. PMID 29256049
- See also: Results available on register — https://www.clinicaltrialsregister.eu/ctr-search/search?query=FLT2504